CLINICAL TRIAL: NCT06762613
Title: Enhancing CBCT-Guided Lung Nodule Puncture Efficiency With Generative AI
Brief Title: Functional Innovation and Application Research of Domestic Advanced Low-Dose DSA/CT-DSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GPS-lung001
Record Dates: First submitted 2024-12-15; First posted 2025-01-07 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Lung Nodules
Keywords: Generative AI; Lung puncture; Cone beam CT; DSA
MeSH Terms: interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPS guided lung puncture (Experimental): Participants will receive percutaneous lung puncture under the guidance of GPS.
  Interventions: Combination Product: Generative AI Based Puncture Surgery Navigation System
- CBCT guided lung puncture (Placebo Comparator): Participants will receive percutaneous lung puncture under the guidance of cone beam CT.
  Interventions: Device: Cone beam CT

INTERVENTIONS:
Combination Product: Generative AI Based Puncture Surgery Navigation System — Participants will receive percutaneous lung puncture under the guidance of GPS.
  Arms: GPS guided lung puncture
Device: Cone beam CT — Participants will receive percutaneous lung puncture under the guidance of cone beam CT.
  Arms: CBCT guided lung puncture

SUMMARY:
The goal of this clinical trial is to learn if Generative AI Based Puncture Surgery Navigation System (GPS) can guide lung puncture in adults better. It will also learn about the quality improvement of cone beam CT (CBCT) by GPS. The main questions it aims to answer are:

* Does GPS lower the number of punctures, radiation dose, and complications of participants undergo percutaneous lung puncture?
* Does GPS improve the quality of CBCT images? Researchers will compare GPS to a conventional CBCT guided percutaneous lung puncture to see if GPS can improve the efficacy of lung puncture.

Participants will:

* Take the percutaneous lung puncture by the guidance of GPS or conventional CBCT (placebo)
* The number of punctures, the success rate of the procedure, the radiation dose, intraoperative complications and postoperative complications at 7 days will be recorded
* The images of CBCT will be collected

ELIGIBILITY:
Inclusion Criteria:

* Participants who require CBCT-guided precutaneous lung puncture (PLP) and meet the clinical indications for the procedure.
* Participants with pre-operation CT images available.
* Participants whose physical condition is suitable for PLP.

Exclusion Criteria:

* Participants have metallic implants in the body, which severely affects the image quality.
* Participants with a history of allergy or serious adverse reactions to iodine contrast media or other related drugs.
* Participants are pregnant or breastfeeding.
* Participants are unwilling or unable to sign informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Number of puncture needles of participants for GPS and CBCT-guided lung puncture procedures. | From enrollment to the end of the lung puncture procedure.
  The number of punctures was defined as the number of punctures performed throughout the percutaneous lung puncture procedure.

SECONDARY OUTCOMES:
Radiation dose for GPS and CBCT-guided lung puncture procedures. | From enrollment to the end of the lung puncture procedure.
  Radiation dose was defined as the radiation dose generated throughout the percutaneous lung puncture procedure.
Puncture time for GPS and CBCT-guided lung puncture procedures. | From enrollment to the end of the lung puncture procedure.
  Puncture time was defined as the duration of the entire percutaneous lung puncture procedure.
Intraoperative and postoperative complications of participants for GPS and CBCT-guided lung puncture procedures. | From enrollment to the end of the lung puncture procedure at 1 week.
  Intraoperative and postoperative complications were defined as those arising in parricipants during percutaneous lung puncture and within 7 days after puncture.

OTHER OUTCOMES:
Algorithmic performance (peak signal-to-noise ratio) | Through study completion, an average of three months.
  peak signal-to-noise ratio (PSNR) is a metric used to measure the quality of an image or video, assessing the degree of distortion by comparing the peak signal power to the mean square error (MSE) between the original signal and the compressed or processed signal. PSNR is measured in decibels (dB), with higher values indicating less distortion and better image or video quality.
Algorithmic performance (structural similarity) | Through study completion, an average of 3 months.
  Structural similarity (SSIM) is a metric for evaluating the similarity of two images. SSIM value is between 0 and 1, the larger the value, the more similar the images are.
Doctors' scoring of image and lesion quality | Through study completion, an average of 3 months.
  Doctors' scoring of image and lesion quality were got based on the 5-point scale Likert (1-5 points). Rated 5 out of 5 for very good images, 4 out of 5 for good, 3 out of 5 for moderate, 2 out of 5 for poor, 1 out of 5 for very poor.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Wuhan Union Hospital, Wuhan, Hubei
  - Wuhan Union Jinyinhu Hospital, Wuhan, Hubei
  - Wuhan Union West Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Deng L, Ji Y, Huang S, Yang X, Wang J. Synthetic CT generation from CBCT using double-chain-CycleGAN. Comput Biol Med. 2023 Jul;161:106889. doi: 10.1016/j.compbiomed.2023.106889. Epub 2023 Apr 3. PMID 37244147
- [Result] Ren Q, Zhou Y, Yan M, Zheng C, Zhou G, Xia X. Imaging-guided percutaneous transthoracic needle biopsy of nodules in the lung base: fluoroscopy CT versus cone-beam CT. Clin Radiol. 2022 May;77(5):e394-e399. doi: 10.1016/j.crad.2022.02.005. Epub 2022 Feb 25. PMID 35227506
- [Result] Choo JY, Park CM, Lee NK, Lee SM, Lee HJ, Goo JM. Percutaneous transthoracic needle biopsy of small (</= 1 cm) lung nodules under C-arm cone-beam CT virtual navigation guidance. Eur Radiol. 2013 Mar;23(3):712-9. doi: 10.1007/s00330-012-2644-6. Epub 2012 Sep 14. PMID 22976917
- [Result] Rotolo N, Floridi C, Imperatori A, Fontana F, Ierardi AM, Mangini M, Arlant V, De Marchi G, Novario R, Dominioni L, Fugazzola C, Carrafiello G. Comparison of cone-beam CT-guided and CT fluoroscopy-guided transthoracic needle biopsy of lung nodules. Eur Radiol. 2016 Feb;26(2):381-9. doi: 10.1007/s00330-015-3861-6. Epub 2015 Jun 6. PMID 26045345
- [Result] Steiling K, Kathuria H, Echieh CP, Ost DE, Rivera MP, Begnaud A, Celedon JC, Charlot M, Dietrick F, Duma N, Fong KM, Ford JG, Gould MK, Holguin F, Perez-Stable EJ, Tanner NT, Thomson CC, Wiener RS, Wisnivesky J. Research Priorities for Interventions to Address Health Disparities in Lung Nodule Management: An Official American Thoracic Society Research Statement. Am J Respir Crit Care Med. 2023 Mar 15;207(6):e31-e46. doi: 10.1164/rccm.202212-2216ST. PMID 36920066
- [Result] Mazzone PJ, Lam L. Evaluating the Patient With a Pulmonary Nodule: A Review. JAMA. 2022 Jan 18;327(3):264-273. doi: 10.1001/jama.2021.24287. PMID 35040882

DOCUMENTS (3):
  • Study Protocol (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT06762613/Prot_003.pdf
  • Statistical Analysis Plan (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT06762613/SAP_004.pdf
  • Informed Consent Form (2024-12-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT06762613/ICF_002.pdf